CLINICAL TRIAL: NCT00939627
Title: Phase II Randomized Trial of the Combination of Cetuximab and Sorafenib or Single Agent Cetuximab in Patients With Refractory, Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Phase II Randomized Trial of the Combination of Cetuximab and Sorafenib or Single Agent Cetuximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02847; NCI-2012-02847 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC-15780 (Other: H. Lee Moffitt Cancer Center and Research Institute); 8070 (Other: CTEP); P30CA076292 (NIH); N01CM00100 (NIH)
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2015-09-01 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Cetuximab; Sorafenib

ARMS (2):
- Arm I (cetuximab and placebo) (Placebo Comparator): Patients receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 and oral placebo twice daily on days 1-21.
  Interventions: Biological: cetuximab; Other: placebo; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment
- Arm II (cetuximab and sorafenib tosylate) (Experimental): Patients receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 and oral sorafenib tosylate twice daily on days 1-21.
  Interventions: Biological: cetuximab; Drug: sorafenib tosylate; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm I (cetuximab and placebo)
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
  Arms: Arm II (cetuximab and sorafenib tosylate)
Other: laboratory biomarker analysis — Correlative studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether cetuximab is more effective when given alone or together with sorafenib tosylate in treating patients with head and neck cancer. This randomized phase II trial is studying cetuximab to see how well it works when given together with or without sorafenib tosylate in treating patients with refractory, recurrent, and/or metastatic head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the progression free survival (PFS) of the combination of cetuximab and sorafenib to that of cetuximab alone in patients with recurrent, refractory or metastatic squamous cell carcinoma of the head and neck (SCCHN).

SECONDARY OBJECTIVES:

I. To evaluate the response rate, overall survival (OS) and toxicity of the combination of cetuximab and sorafenib and of cetuximab alone.

II. To evaluate the presence of EGFRvIII mutation, increased EGFR gene copy number and activated EGFR gene expression signature, and correlate with clinical parameters (RR, OS and PFS) in the cetuximab alone and cetuximab/sorafenib arms.

III. To evaluate whether VEGF receptor family and their ligand expression can predict response to cetuximab/sorafenib.

IV. To determine the proteomic profiles in serum and tumors that can predict the response and survival upon the treatment with cetuximab or cetuximab/sorafenib.

V. To evaluate the effect of therapy on both general and head and neck specific functionality, symptom burden and QOL.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 and oral placebo twice daily on days 1-21. (oral placebo closed as of 02/18/2010).

ARM II: Patients receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 and oral sorafenib tosylate twice daily on days 1-21.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Paraffin embedded tissue samples are collected at baseline for pharmacogenomic studies and blood samples are collected at baseline and for the first 3 courses for research purposes. Quality of life and symptom burden are assessed by Vanderbilt Head and Neck Symptom Survey, FACT-HN, and Fatigue and Pain Inventory questionnaires at baseline, at day 43, and at 3 and 6 months.

After completion of study treatment, patients are followed periodically for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent, refractory or metastatic squamous cell carcinoma of oral cavity, oropharynx and larynx, hypopharynx or paranasal sinus, head and neck unknown primary or nasopharyngeal carcinoma WHO type 1; patients with recurrent, refractory or metastatic squamous cell carcinoma of oral cavity, oropharynx and larynx, hypopharynx or paranasal sinus, head and neck unknown primary or nasopharyngeal carcinoma WHO type 1; patients may have had up to 1 prior palliative chemotherapy for recurrent or metastatic disease; please note that chemotherapy given as part of a regimen for curative intent for recurrent disease does not count as "prior chemotherapy;" patients must not presently be candidates for curative therapy
* ECOG performance status 0, 1 or 2
* Hemoglobin >= 9.0/dl
* Absolute-neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 x ULN
* ALT and AST =< 2.5 x ULN (=< 5 x ULN for patients with liver involvement)
* INR < 1.5 or a PT and PTT within normal limits
* Creatinine =< 1.5 x ULN
* If primary therapy was given for curative intent, at least 4 weeks must have elapsed after completion of primary therapy prior to enrollment on this clinical trial; however, toxicities from prior treatment must have resolved to grade 1 or less
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of the treatment; women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation (i.e, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and for a minimum of 3 months following the last dose of chemotherapy; male subject agrees to use an acceptable method for contraception for the duration of the study and for a minimum of 3 months following the last dose of chemotherapy
* Patients must have a measurable disease defined by RECIST criteria
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care; patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial

Exclusion Criteria:

* Prior treatment with sorafenib or cetuximab
* Patients with active clinically significant infection or with a fever >= 38.5º C within 3 days of the first scheduled day of protocol treatment
* History of prior malignancy within the past 3 years except for curatively treated basal cell carcinoma and squamous cell carcinoma of the skin, CIN or localized prostate cancer with a current PSA < 1.0 mg/dL on 2 successive evaluations at least 3 months apart, with the most recent evaluation within 4 weeks of study entry
* Patients with known hypersensitivity to sorafenib or cetuximab
* Prior severe infusion reaction to a monoclonal antibody
* History of hand-foot syndrome
* Pregnant or lactating; sexually active women of childbearing potential must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized
* Known untreated brain metastasis; patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis or progression of brain metastasis; patients with treated brain metastasis are eligible for study as long as no evidence of progression of CNS disease; hemorrhagic brain metastases are not allowed on study
* Uncontrolled comorbid illness
* Patients with HIV who are taking antiretroviral mediations will be excluded because of the potential interactions of anti-retroviral medications with these agent; however, given the potential immune modulating effects of sorafenib, investigators should still be very cautious about placing HIV positive patients on this trial as the effects of these medications on the HIV virus itself are not know
* History of allogeneic transplant
* Patient has received other investigational drugs within 28 days before enrollment
* Cardiac disease: congestive heart failure > class II NYHA; patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months; significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension (defined as defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction will also be excluded from study; cardiac ventricular arrhythmias requiring anti-arrhythmic therapy will also be excluded from study
* Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event > CTCAE grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event > CTCAE grade 3 within 4 weeks of first dose of study drug
* Tumor that invades the carotid artery as shown unequivocally by imaging studies
* Serious non-healing wound, ulcer, or bone fracture
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug
* Use of St. John's Wort or rifampin (rifampicin)
* Use of the following medications will not be allowed within 4 weeks prior to enrollment on the study and during the study: ketoconazole, itraconazole, ritonavir, cyclosporine, carbamazepine, phenytoin, phenobarbital; products containing grapefruit juice will not be allowed while on study
* Known or suspected allergy to sorafenib or any agent given in the course of this trial
* Any malabsorption problem
* Known HIV positive patients will be excluded from trial due to the potential immune modulation that these agents may cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Gilbert, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (8):
- United States (8):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Billings Clinic, Billings, Montana
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Southeast Phase II Consortium (SEP2C) study enrolling participants at seven participating sites during August 2009 through October 2011.
Pre-assignment Details: Fifty-five patients were consented and assigned to a treatment arm; 3 withdrew before treatment. Fifty-two patients were treated on study. After 19 patients were enrolled, the trial was amended to remove the placebo (and blinding) due to issues with placebo tablet solubility.
Groups:
- Arm A - Cetuximab: Patients were to receive cetuximab 400 mg/m^2 IV over 60-120 minutes on days 1, 8, and 15 and oral placebo twice daily on days 1-21. After 19 patients were enrolled, the trial was amended to remove the placebo (and blinding) due to issues with placebo tablet solubility..
- Arm B - Cetuximab and Sorafenib Tosylate: Patients received cetuximab 400 mg/m^2 IV over 60-120 minutes on days 1, 8, and 15 and oral sorafenib tosylate 400 mg by mouth twice daily on days 1-21.
- Participants Who Did Not Receive Treatment.: Placebo Arm: The protocol was amended and this arm was removed.
Period: Overall Study
Arm/Group | Arm A - Cetuximab | Arm B - Cetuximab and Sorafenib Tosylate | Participants Who Did Not Receive Treatment.
Started | 27 | 28 | 0
Completed | 0 | 0 | 0
Not Completed | 27 | 28 | 0
Not completed — Disease Progression | 16 | 12 | 0
Not completed — Adverse Event | 6 | 7 | 0
Not completed — Death | 0 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 0
Not completed — Other complicating disease | 1 | 1 | 0
Not completed — Not compliant | 2 | 0 | 0
Not completed — No off-tx reason given | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline participant measures are based on total eligible, consented, patients. Three of 55 consenting patients did not receive treatment. One patient had disease progression before treatment and 2 patients withdrew before treatment, resulting in 52 patients on treatment.
Groups:
- Arm A - Cetuximab: Patients were to receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 and oral placebo twice daily on days 1-21. After 19 patients were enrolled, the trial was amended to remove the placebo (and blinding) due to issues with placebo tablet solubility.
- Arm B - Cetuximab and Sorafenib Tosylate: Patients receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 and oral sorafenib tosylate twice daily on days 1-21.
- Total: Total of all reporting groups
Arm/Group | Arm A - Cetuximab | Arm B - Cetuximab and Sorafenib Tosylate | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 7 | 7 | 14
Age, Customized [Median (Full Range); unit: years] | 59 [26 to 74] | 60 [42 to 71] | 59 [26 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 25 | 23 | 48
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Estimated probable duration of life without disease progression, from on-study date to earlier of progression date or date of death from any cause, using the Kaplan-Meier method with censoring (see analysis population description for additional details). Disease progression is defined under Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as >=20% increase in sum of longest diameters of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions.
Time Frame: On-study date to lesser of date of progression or date of death from any cause (assessed up to 3 years)
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where either death or progression is an event, with censoring for non-progressed, non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Cetuximab | Arm B - Cetuximab and Sorafenib Tosylate
Number analyzed (Participants) | 26 | 26
months | 3 [1.9 to 5.0] | 3.2 [1.8 to 4.2]

2. Secondary Outcome: Best Response
Description: Number of patients in each response category, per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, summarized as follows for target lesion criteria (see RECIST v1.1 for additional details): complete response (CR),disappearance of target lesions; partial response (PR), >=30% decrease in sum of longest diameter of target lesions; progressive disease (PD), >=20% increase in sum of longest diameter (LD) of target lesions or appearance of new lesions; stable disease (SD), insufficient change in target lesions or new lesions to qualify as either PD or SD.
  Patients are categorized according to the best response achieved prior to occurrence of progressive disease, where best response hierarchy is CR>PR>SD>PD.
Time Frame: On-treatment date to date of disease progression (assessed up to 3 years)
Population: All patients with best overall response data. Patients are excluded if best overall response data is missing or if the patient is not evaluable for best overall response.
Measure: Number; unit: participants
Arm/Group | Arm A - Cetuximab | Arm B - Cetuximab and Sorafenib Tosylate
Number analyzed (Participants) | 22 | 20
participants
  Patients with Complete Response | 0 | 0
  Patients with Partial Response | 1 | 2
  Patients with Stable Disease | 11 | 10
  Patients with Progressive Disease | 9 | 8
  Patients Not Evaluable | 4 | 6
  Patients with Less Than Partial Response | 1 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Estimated probable duration of life from on-study date to date of death from any cause, using the Kaplan-Meier method with censoring (see analysis population description for additional details)
Time Frame: On-study date to date of death from any cause (assessed up to 3 years)
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where death is an event, with censoring for non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Cetuximab | Arm B - Cetuximab and Sorafenib Tosylate
Number analyzed (Participants) | 26 | 26
months | 9 [5.2 to 12.9] | 5.7 [4.2 to 10.8]

4. Secondary Outcome: Number of Participants With Each Worst-Grade Toxicity
Description: Count of patients according to the worst-grade toxicity experienced by each, where worst-grade toxicity is per NCI common toxicity criteria: grade 1, mild; grade 2, moderate; grade 3, severe; grade 4, life-threatening; grade 5, death
Time Frame: On-study date to 30 days following final dose of study drug
Population: Total number of patients reported with any toxicity. Because not all patients experience a toxicity, and some experience more than one; the number of patients analyzed does not coincide with the number of patients on study.
Measure: Number; unit: participants
Arm/Group | Arm A - Cetuximab | Arm B - Cetuximab and Sorafenib Tosylate
Number analyzed (Participants) | 23 | 24
participants
  Number of Patients with Worst-Grade Toxicity 1 | 6 | 7
  Number of Patients with Worst-Grade Toxicity 2 | 11 | 4
  Number of Patients with Worst-Grade Toxicity 3 | 5 | 12
  Number of Patients with Worst-Grade Toxicity 4 | 1 | 1
  Number of Patients with Worst-Grade Toxicity 5 | 0 | 0

5. Secondary Outcome: Gene Expression Levels
Description: Formalin-fixed, paraffin-embedded (FFPE) tumors were collected. The FFPE tumors were to be evaluated for p16 expression using immunohistochemistry staining with antibody. Gene Expression Levels (positive when >70% cells stained, otherwise negative) were to be described using frequencies.
Time Frame: Pre-therapy
Population: Due to an insufficient amount of tumor tissue available to complete planned analysis, this analysis was abandoned.
Arm/Group | Arm A - Cetuximab | Arm B - Cetuximab and Sorafenib Tosylate
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Survival Associated With Immunomodulatory Cytokines
Description: Twelve immunomodulatory cytokines were selected based on previous a feasibility study and detected using multiplex Luminex bead assays from patient's plasma. One cytokines, HGF, was eliminated due to extremely low expression. Three representative cytokines, TGF-beta 1, IL-8 and VEGF were to be evaluated for association with survival due to clustering.
Time Frame: Pre-therapy, up to about 42 months (follow-up for overall survival)
Population: Data were not collected due to an insufficient amount of tumor tissue available.
Arm/Group | Arm A - Cetuximab | Arm B - Cetuximab and Sorafenib Tosylate
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Quality of Life
Description: Quality of Life Survey results.
Time Frame: up to 3 years
Population: Data were not collected as The Quality of Life survey instrument was not completed by study participants..
Arm/Group | Arm A - Cetuximab | Arm B - Cetuximab and Sorafenib Tosylate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years, 4 months
Description: All participants who received treatment.
Groups:
- Arm B - Cetuximab and Sorafenib Tosylate: Patients received cetuximab IV over 60-120 minutes on days 1, 8, and 15 and oral sorafenib tosylate twice daily on days 1-21.
Arm/Group | Arm A - Cetuximab | Arm B - Cetuximab and Sorafenib Tosylate
Serious Adverse Events (participants affected / at risk) | 5/26 | 10/27
Other Adverse Events (participants affected / at risk) | 25/26 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Cetuximab (N=26) | Arm B - Cetuximab and Sorafenib Tosylate (N=27)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Death NOS (General disorders) | 1 (1) | 3 (3)
Infusion related reaction (General disorders) | 0 (0) | 1 (2)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
Nervous system disorders - Other - related to pain meds (Psychiatric disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Cetuximab (N=26) | Arm B - Cetuximab and Sorafenib Tosylate (N=27)
Fatigue (General disorders) | 19 (31) | 18 (27)
Pain (General disorders) | 4 (5) | 6 (7)
Chills (General disorders) | 2 (2) | 2 (2)
Edema - limbs (General disorders) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (11) | 8 (8)
Nausea (Gastrointestinal disorders) | 7 (11) | 7 (11)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 10 (14)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 5 (7)
Mucositis oral (Gastrointestinal disorders) | 4 (5) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 5 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 1 (1) | 2 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (21) | 10 (18)
Rash acneiform (Skin and subcutaneous tissue disorders) | 9 (12) | 9 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
Skin and subcutaneous tissue disorders - other (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 6 (7) | 8 (11)
Hyponatremia (Metabolism and nutrition disorders) | 4 (5) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (7) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (8) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (6) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 11 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (10)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 6 (8) | 8 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 1 (1)
Weight loss (Investigations) | 3 (4) | 6 (7)
Alkaline phosphatase increased (Investigations) | 3 (5) | 3 (3)
Skin infection (Infections and infestations) | 4 (4) | 0 (0)
Infections and infestations - other (Infections and infestations) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
Eye disorders - Other (Eye disorders) | 5 (5) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 2 (4) | 2 (3)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (8)
Leukocytosis (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 3 (3)
Anaphylaxis (Immune system disorders) | 1 (1) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (4)
Tinnitus (Ear and labyrinth disorders) | 2 (3) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) | 1 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Muscoloskeletal and connective tissue disorders - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Immune system disorders - Other (Immune system disorders) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (3) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Psychiatric disorders - Other (Psychiatric disorders) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Hemoglobin increased (Investigations) | 1 (3) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (2)
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (2)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
General disorders and administration site conditions (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Accrual ended early based on planned interim analysis, but the study was completed with existing participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less